CLINICAL TRIAL: NCT05118997
Title: Active Removal of IntraCerebral Hematoma Via Active Irrigation of the Ventricular System
Brief Title: Active Removal of IntraCerebral Hematoma Via Active Irrigation
Acronym: ARCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRRAS (Industry)
Collaborators: University of Helsinki (Other); Northwestern University (Other); West Virginia University (Other); Klinikum Bergmannstrost (Unknown); Stony Brook University Hospital (Unknown); Icahn School of Medicine at Mount Sinai (Other); Buffalo General Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2021-10-15; First posted 2021-11-12 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Hemorrhage; Intraventricular Hemorrhage
Keywords: Hemorrhage; Cerebral Hemorrhage; Intraventricular Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Arm #1 (Experimental): IRRAflow with manual tPA administration followed by Active Fluid Exchange
  Interventions: Device: IRRAflow
- Treatment Arm #2 (Experimental): IRRAflow with continuous infusion of tPA combined with Active Fluid Exchange
  Interventions: Device: IRRAflow
- Treatment Arm #3 (Active Comparator): Standard EVD with manual tPA administration
  Interventions: Device: EVD

INTERVENTIONS:
Device: IRRAflow — IRRAflow consists of a control unit and disposables (dual-lumen catheter and tube set) to offer an integrated and synchronized active fluid exchange system. Active fluid exchange is the combination of traditional gravity-driven drainage with periodic, controlled irrigation of the catheter probe to exchange any pathological fluid collection with neutral physiological fluids.
  Arms: Treatment Arm #1; Treatment Arm #2
Device: EVD — An external ventricular drain (EVD), also known as a ventriculostomy or extraventricular drain, is a device used in neurosurgery to treat hydrocephalus and relieve elevated intracranial pressure when the normal flow of cerebrospinal fluid inside the brain is obstructed.
  Arms: Treatment Arm #3

SUMMARY:
Study evaluating if active irrigation by IRRAflow® with infusion of tPA will reduce the time needed for clearance of intracerebral and intraventricular hemorrhage compared with passive drainage.

DETAILED DESCRIPTION:
The ARCH study is an international prospective, controlled, randomized, multicenter study to evaluate the hypothesis that active irrigation with IRRAflow® will reduce the time needed for clearance of intraventricular and intracerebral blood from intraventricular and intracerebral space compared with passive drainage and administration of tPA. This might affect the patient neurological outcome assessed by GCS and mRankin scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Need of EVD
3. Active treatment
4. Signed informed consent obtained

   a. Based on institutional and country laws
5. Spontaneous ICH with maximum 30 square cm's
6. If needed, normal coagulation profile (PT, PTT, platelet count)
7. Treatment within 72 hours of ictus
8. Ability to administer 2.0 mg of tPA per day for 3 days

Exclusion Criteria:

1. Age < 18 years
2. No need of EVD
3. Patient has fixed and dilated pupils
4. Coagulopathy uncorrectable
5. Vascular pathology (e.g. Aneurysm involvement, AVM involvement)
6. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of evacuation of intraventricular hematoma by Active External Ventricular Drainage (IRRAflow) with tPA administration compared to Passive External Ventricular Drainage (EVD) with tPA administration. | Intra-procedure
  Efficacy is defined as the efficiency of each arm to remove the hematoma (70% cm3). Safety is measured as the frequency of bacterial central nervous system (measures as positive bacterial growth in cerebrospinal fluid), symptomatic brain bleeds (clinical symptoms drop in modified Rankin scale), and mortality (death).
Radiographic evaluation of ventricular blood removal as measured by head CT scan | Intra-procedure
  Change in blood volume (cm3) measured between stability scan and end of treatment scan.
Comparison of patient outcome between groups at as measured by the Glasgow Coma Scale, extended Glasgow Outcome Scale, modified Rankin Scale. | 0-30 days post discharge from hospital
  Defined as the comparison of patients outcomes between the three groups as measured by Glasgow Coma Scale, extended Glasgow Outcome Scale, and modified Rankin Scale.

SECONDARY OUTCOMES:
Procedural Success | Intra-Procedural
  Less than or equal to 30% residual clot burden in the ventricular system
Technical Success | Intra-Procedural
  Percentage of patients in which correct placement of IRRAflow and EVD catheter occurred
Technical Success | Intra-Procedural
  Percent obstruction of the IRRAflow catheter and EVD catheter
Safety - Catheter misplacement | Intra-Procedural
  Measurement of if the catheter needs to be re-inserted or re-positioned.
Safety - Infection | Intra-Procedural
  Comparison of rate of infection as measured by routine cerebrospinal fluid (CSF) analysis
Safety - Bleeding events | Intra-Procedural
  Comparison of new bleeding events on routine neuroimaging

OTHER OUTCOMES:
Length of ICU stay (days) | Intra-Procedural
  Time (days) the patient is admitted to the ICU till the patient is discharged from the ICU
Length of overall length (days) of hospital stay | Intra-Procedural
  Time (days) the patient is admitted to the hospital till the patient is discharged from the hospital
Rate of mortality during treatment | Intra-Procedural
  Percentage of patients having a mortality event during active treatment
Rate of shunt dependency | 30 days
  Percentage of patients that require a shunt after treatment
Radiological evaluation of ventricles as measured by CT scan of head | Intra-Procedural
  Radiologic evaluation of the ventricles by the neurosurgeon or radiologist
Duration of EVD and IRRAflow catheter in place | Intra-Procedural
  Number of days between catheter insertion and with drawl of the catheter
Rate of clot removal as assessed by CT | Intra-Procedural
  Change in blood volume measured between stability scan and end of treatment scan
Duration of catheter drainage | Intra-Procedural
  Number of days catheter was utilized for drainage
Catheter occlusion rate | Intra-Procedural
  Percentage of time in which the catheter is unable to drain
Revision rate of the EVD and IRRAflow catheter | Intra-Procedural
  Percentage of time that the physician must replace or manipulate the EVD or IRRAflow catheter
Repeat hemorrhagic events | Intra-Procedural
  Number of repeated symptomatic hemorrhagic events
Catheter occlusion | Intra-Procedural
  Number of flushes required to clear a catheter occlusion
Functional Status | Intra-Procedural
  modified Rankin Score (mRS)
Functional Status | 30 day
  Difference in modified Rankin Score (mRS) as proportioned to IVH size
Total cost of procedure | Intra-Procedural
  Measured as total cost involved in treating patient during treatment with IRRAflow and EVD

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Rezai Jahromi, MD, Principal Investigator — University of Helsinki; Babak Jahromi, MD, Principal Investigator — Northwestern University
Locations (1):
- Helsinki University, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajjoub K, Hess RM, O'Connor TE, Khan A, Siddiqui AH, Levy EI. Drainage, Irrigation, and Fibrinolytic Therapy (DRIFT) for Adult Intraventricular Hemorrhage Using IRRAflow(R) Self-Irrigating Catheter. Cureus. 2021 May 22;13(5):e15167. doi: 10.7759/cureus.15167. PMID 34168930
- [Background] Qureshi AI, Mendelow AD, Hanley DF. Intracerebral haemorrhage. Lancet. 2009 May 9;373(9675):1632-44. doi: 10.1016/S0140-6736(09)60371-8. PMID 19427958
- [Background] Qureshi AI, Tuhrim S, Broderick JP, Batjer HH, Hondo H, Hanley DF. Spontaneous intracerebral hemorrhage. N Engl J Med. 2001 May 10;344(19):1450-60. doi: 10.1056/NEJM200105103441907. No abstract available. PMID 11346811
- [Background] Sacco S, Marini C, Toni D, Olivieri L, Carolei A. Incidence and 10-year survival of intracerebral hemorrhage in a population-based registry. Stroke. 2009 Feb;40(2):394-9. doi: 10.1161/STROKEAHA.108.523209. Epub 2008 Nov 26. PMID 19038914
- [Background] Findlay JM, Weir BK, Gordon P, Grace M, Baughman R. Safety and efficacy of intrathecal thrombolytic therapy in a primate model of cerebral vasospasm. Neurosurgery. 1989 Apr;24(4):491-8. doi: 10.1227/00006123-198904000-00002. PMID 2496328
- [Background] Pang D, Sclabassi RJ, Horton JA. Lysis of intraventricular blood clot with urokinase in a canine model: Part 2. In vivo safety study of intraventricular urokinase. Neurosurgery. 1986 Oct;19(4):547-52. doi: 10.1227/00006123-198610000-00009. PMID 3491339
- [Background] Davis SM, Broderick J, Hennerici M, Brun NC, Diringer MN, Mayer SA, Begtrup K, Steiner T; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Hematoma growth is a determinant of mortality and poor outcome after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1175-81. doi: 10.1212/01.wnl.0000208408.98482.99. PMID 16636233
- [Background] Steiner T, Diringer MN, Schneider D, Mayer SA, Begtrup K, Broderick J, Skolnick BE, Davis SM. Dynamics of intraventricular hemorrhage in patients with spontaneous intracerebral hemorrhage: risk factors, clinical impact, and effect of hemostatic therapy with recombinant activated factor VII. Neurosurgery. 2006 Oct;59(4):767-73; discussion 773-4. doi: 10.1227/01.NEU.0000232837.34992.32. PMID 17038942